CLINICAL TRIAL: NCT04975828
Title: Correlation Between Micro Vascular Complications and Severity of Coronary Artery Disease in Type 2 DM
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Islam Khaled Fathy, resident at internal medicine, Sohag University
Other Study IDs: Soh-Med-21-07-02
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Patients With Type 2 DM Who Underwent Coronary Angiography Due to Coronary Artery Disease and Presence of Microvascular Complications in Same Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- patients type 2 DM with coronary artery disease and diabetic retinopathy.
  Interventions: Diagnostic Test: albumin creatinine ratio -EGFR-fundus examination- coronary angiography.
- patients type 2 DM with coronary artery disease and diabetic neuropathy.
  Interventions: Diagnostic Test: albumin creatinine ratio -EGFR-fundus examination- coronary angiography.
- patients type 2 DM with coronary artery disease and diabetic nephropathy
  Interventions: Diagnostic Test: albumin creatinine ratio -EGFR-fundus examination- coronary angiography.
- patient type 2 DM with coronary artery disease and non microvascular complications.
  Interventions: Diagnostic Test: albumin creatinine ratio -EGFR-fundus examination- coronary angiography.

INTERVENTIONS:
Diagnostic Test: albumin creatinine ratio -EGFR-fundus examination- coronary angiography. — albumin creatinine ratio and EGFR to assess. diabetic nephropathy. fundus examination to assess. diabetic retinopathy. assess of coronary artery disease by coronary angiography. assess diabetic nephropathy by neurologic examination.

SUMMARY:
Diabetes is a major cause of morbidity and mortality worldwide and it contributes substantially to healthcare costs. Type 2 Diabetes mellitus is the most common type of diabetes accounting for approximately (90%) of all cases.

Type 2 DM carries a two to six times risk of death from cardiovascular etiologies, such that age adjusted prevalence of white Americans for coronary artery disease (CAD) is double in those with type 2 DM than those without .

ELIGIBILITY:
Inclusion Criteria:

100 Cases were selected with type II (DM) patients who had been admitted for coronary angiography because of suspected (CAD) to the Catheter lab unit of Sohag University Hospital.

Exclusion Criteria:

1. Type 1 DM.
2. Smoker.
3. Hypertension.
4. Pregnant women.
5. Patient known non diabetic retinal disease non diabetic. nephropathy or neuropathy.
6. History of familial dyslipidemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled 100 patients known type 2 DM with coronary artery disease and coronary angiography done to diagnosis coronary artery disease then assess microvascular complications in those patients by fundus examination-neurologic examination-albumin creatinine ratio-EGFR. IN STUDY investigator exclude any other cause can lead to microvascular complications example hypertension.
  aim of study to early predict coronary artery disease in patient with type 2 DM if microvascular complication presenet by non invasive investigation as stress ECG.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
correlation between microvascular complications and severity of coronary disease in type2 DM. | 4 months
  outcome of study to assess correlation between coronary artery disease and microvascular complications in type 2 DM to early predict coronary artery disease in patient type 2 DM with microvascular complications by non invasive methods as stress ECG or CT coronary angio or cardiac MRI and prevent serious complications as myocardial infarction.
  assess microvascular complication as follow albumin creatinine ratio and EGFR to assess. diabetic nephropathy. fundus examination to assess. diabetic retinopathy. assess of coronary artery disease by coronary angiography. assess diabetic nephropathy by neurologic examination.

CONTACTS AND LOCATIONS:
Locations (1):
- Osama R Elsherief, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ybarra-Munoz J, Jurado-Campos J, Garcia-Gil M, Zabaleta-Del-Olmo E, Mir-Coll T, Zabalegui A, Vidal J, Romeo JH. Cardiovascular disease predicts diabetic peripheral polyneuropathy in subjects with type 2 diabetes: A 10-year prospective study. Eur J Cardiovasc Nurs. 2016 Jun;15(4):248-54. doi: 10.1177/1474515114565215. Epub 2014 Dec 19. PMID 25527522
- [Background] Dal Canto E, Ceriello A, Ryden L, Ferrini M, Hansen TB, Schnell O, Standl E, Beulens JW. Diabetes as a cardiovascular risk factor: An overview of global trends of macro and micro vascular complications. Eur J Prev Cardiol. 2019 Dec;26(2_suppl):25-32. doi: 10.1177/2047487319878371. Epub 2019 Nov 13. PMID 31722562
- [Background] Glovaci D, Fan W, Wong ND. Epidemiology of Diabetes Mellitus and Cardiovascular Disease. Curr Cardiol Rep. 2019 Mar 4;21(4):21. doi: 10.1007/s11886-019-1107-y. PMID 30828746